CLINICAL TRIAL: NCT05034211
Title: A Comparison Between 2 Methods of Local Anesthetic Administration for Maintaining Labor Analgesia After Dural Puncture Epidural
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieio Hospital (Other)
Responsible Party: Principal Investigator, Polyxeni Theodosopoulou, Resident anesthesiologist, Aretaieio Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 342/25/5/21
Record Dates: First submitted 2021-06-15; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Labor Pain; Epidural; Pain, Labor
Keywords: dural puncture; programmed intermittent bolus; labor analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Programmed intermittent Bolus Epidural technique (Active Comparator): 10ml ropivacaine 0,2% and 1,5 mcg/ml fentanyl, will be administered every 60 minutes via an epidural catheter placed for labor analgesia on L2-L3/L3-L4 level
  Interventions: Procedure: Programmed intermittent bolus epidural
- Provider administered bolus epidural technique on patient request (Active Comparator): 10ml ropivacaine 0,2% and 1,5 mcg/ml fentanyl, will be administered by the provider on patient request
  Interventions: Procedure: Provider administered analgesia on patient request

INTERVENTIONS:
Procedure: Programmed intermittent bolus epidural — one arm will receive programmed intermittent boluses of local anesthetic via the epidural catheter on fixed time intervals. Standard 27G Tuohy needle epidural set with epidural catheter insertion on L2-L3 site, with the patient either sitting or in the lateral decubitus position will be used. Local injection with 6 ml lidocaine 2% will be performed before the insertion of the epidural needle
  Arms: Programmed intermittent Bolus Epidural technique
Procedure: Provider administered analgesia on patient request — one arm will receive bolus of local anesthetic via the catheter upon patient request. Standard 27G Tuohy needle epidural set with epidural catheter insertion on L2-L3 site, with the patient either sitting or in the lateral decubitus position will be used. Local injection with 6 ml lidocaine 2% will be performed before the insertion of the epidural needle
  Arms: Provider administered bolus epidural technique on patient request

SUMMARY:
Intermittent epidural bolus technique opens a new era of interest for maintaining labor anlagesia. The study examines programmed intermittent epidural bolus technique on a scheduled basis to provider-administered bolus anlgesia on patient request, after a dural puncture epidural technique.

DETAILED DESCRIPTION:
After dural puncture, an epidural catheter will be placed on nulliparous women between 38 and 40 weeks of gestation presenting for labor . All will receive an test dose of 3ml lidocaine 2%, for properly checking the catheter placement and then an initial dose of 10ml ropivacaine 0,2% with 2 mcg/ml fentanyl. After that, women will be randomly assigned on two groups. Both groups will be receiving the same dose of analgesia (10ml ropivacaine 0,2% plus 1,5 mcg/ml fentanyl. However, one group will be receiving them on scheduled time intervals as programmed intermittent boluses every 60minutes and the other only on patient request for pain relief.

Pain scores, satisfaction, time for adequate analgesia, bromage scores,apgar scores, fetal arterial blood gases, time for delivery and type of delivery will be studied

ELIGIBILITY:
Inclusion Criteria:

-nulliparous women

* 38th week of gestation

Exclusion Criteria:

* patient refusal to have an epidural
* patient refusal to participate
* contraindication for epidural
* ASA>3
* neurologic deficit/impairment
* allergy on local anesthetic chronic pain syndromes

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Total local anesthetic and opioid administration | 24hours
  the total mg of local anesthetic and opioid consumed via the epidural catheter until the neonate delivery

SECONDARY OUTCOMES:
time needed for delivery | 24hours
  how long will it take for the baby to be delivered(in minutes)
total patient satisfaction | 24hours
  from a scale of 0 to 10, higher score signifies better outcome
apgar score | 24hours
  a test given to newborns soon after birth. This test checks a baby's heart rate, muscle tone, and other signs to see if extra medical care or emergency care is needed. The test is usually given twice: once at 1 minute after birth, and again at 5 minutes after birth.The higher the score the better the baby's condition willl be (the scale is from 0 to 10)
Bromage score | 24hours
  This scale assesses the intensity of motor block by the patient's ability to move their lower extremities. O signifies free movement and 4 complete paralysis(higher score means worse outcome)
type of delivery | 24hours
  whether it will be vaginal delivery, vaginal assisted delivery with instruments or a cesarean section
neonatal arterial blood gases | 24hours
  when the baby will be delivered, a neonatal arterial blood gas will be measured
time for sucessful level of analgesia | 24hours
  the time needed after epidural bolus to reach a scale below 3 on the NRS scale for pain assesment
Pain score(NRS scale) | 24hours
  n a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 . O represents no pain and 10 the worst pain ever possible

CONTACTS AND LOCATIONS:
Locations (1):
- Aretaieio Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided